CLINICAL TRIAL: NCT02969889
Title: Intubation in Morbidly Obese: a Comparison of Airtraq and ILMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Zehra Ipek ARSLAN, Assistant Professor, Kocaeli University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: KOU KAEK 2014/137
Record Dates: First submitted 2016-11-18; First posted 2016-11-21 (Estimated); Last update posted 2017-02-03 (Estimated); Status verified 2017-02

CONDITIONS: Intubation; Difficult or Failed; Intubation Complication
Keywords: Airtraq; Intubating laryngeal mask airway; BMI>35

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- intubation time (Active Comparator): handling the device till the endotracheal tube passing through the glottis
  Interventions: Device: Airtraq; Device: ILMA
- insertion time (Active Comparator): handling of the device till the glottic visualization
  Interventions: Device: Airtraq; Device: ILMA

INTERVENTIONS:
Device: Airtraq — video laryngoscope with a channel
Device: ILMA
  Other Names: intubating laryngeal mask airway

SUMMARY:
bmı > 35 morbidly obese patients requiring endotracheal intubation enrolled in this trial. Divided into two groups Airtraq and ILMA. their effectiveness is evaluated.

DETAILED DESCRIPTION:
80 patients, 18-65 years of aged ASA I-III, BMI> 35 patients enrolled in this trial.

Divided into two groups ; Airtraq and ILMA .

BMI>35, upper airway tumour , respiratory infection less than ten days, excluded from this study.

patients demographic and airway variables were recoded. Patients were premedicated. After standard anesthesia induction, anesthesia was induced with propofol and fentanyl. Rocuronium was used for neuromuscular blockade.

The device insertion and intubation times, number of intubation attempts, mucosal damage, need for optimization maneuvers, effects on hemodynamic parameters and postoperative minor complications were recorded.

ELIGIBILITY:
Inclusion Criteria:18-65 years of age

* ASA I-III
* BMI>35

Exclusion Criteria:BMI<35

* patients have airway tumor
* patients undergoing head and neck surgery
* upper respiratory infection less than 10 days prior the surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
intubation time | 1 minute
  handling of the device till the endotracheal tube entering the glottis

CONTACTS AND LOCATIONS:
Overall Officials: Zehra Arslan, Principal Investigator — Kocaeli University Medical Faculty
Locations (1):
- Kocaeli University School of Medicine, Kocaeli, Turkey (Türkiye)